CLINICAL TRIAL: NCT04997902
Title: A Phase 1/2 Open-label, Biomarker-defined Cohort Trial to Evaluate the Safety, Determine the Recommended Combination Dosing, and Assess Early Antitumor Activity of Tipifarnib and Alpelisib for the Treatment of Adult Participants Who Have HRAS-overexpressing and/or PIK3CA-mutated and/or - Amplified Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Combination Trial of Tipifarnib and Alpelisib in Adult Recurrent/ Metastatic Head and Neck Squamous Cell Carcinoma (R/M HNSCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KO-TIP-013
Expanded Access: NCT04809233 (Available)
Record Dates: First submitted 2021-07-27; First posted 2021-08-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: HNSCC
Keywords: HRAS; PIK3CA; PI3K; Tipifarnib; Alpelisib; R/M HNSCC (Recurrent/metastatic Head and Neck Squamous Cell Carcinoma); Head and Neck Cancer; SCCHN
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Hereditary Sensory and Autonomic Neuropathies; Recurrence; Head and Neck Neoplasms | interventions — tipifarnib; Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PIK3CA-dependent (Cohort 1) (Experimental): Adult participants with R/M HNSCC whose tumors harbor PI3KCA (activating) mutations and/or amplifications
  Interventions: Drug: Tipifarnib; Drug: Alpelisib
- HRAS-dependent (Cohort 2) (Experimental): Adult participants with R/M HNSCC whose tumors have increased HRAS dependency, defined as HRAS overexpression
  Interventions: Drug: Tipifarnib; Drug: Alpelisib

INTERVENTIONS:
Drug: Tipifarnib — Oral administration
Drug: Alpelisib — Oral administration
  Other Names: BYL719

SUMMARY:
This phase 1/2 combination trial of tipifarnib, a farnesyltransferase inhibitor, and alpelisib, a PI3K inhibitor in participants with recurrent/metastatic head and neck squamous cell carcinoma (HNSCC) whose tumors overexpress the HRAS protein and/or are PIK3CA-mutated and/or PIK3CA-amplified.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Histologically confirmed head and neck cancer of squamous histology not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
3. Documented treatment failure from at least 1 prior systemic therapy in the R/M setting, unless determined not appropriate.
4. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
5. Has a tumor that is dependent upon HRAS and/or PIK3CA.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
7. Acceptable liver, renal, endocrine, and hematologic function.
8. Must be able to swallow alpelisib whole tablet or oral suspension containing crushed tablets. Feeding tube may not be used for alpelisib administration.
9. Other protocol defined inclusion criteria may apply.

Exclusion Criteria:

1. Histologically confirmed salivary gland, thyroid, (primary) cutaneous squamous or nonsquamous histologies (eg, mucosal melanoma).
2. Ongoing treatment with certain anticancer agents.
3. Prior treatment (at least 1 full treatment cycle) with an FTI or PI3K, mTOR, or AKT inhibitor.
4. Received treatment for unstable angina, myocardial infarction, and/or cerebro-vascular attack within the prior 6 months.
5. Non-tolerable Grade 2, or ≥ Grade 3 neuropathy or evidence of unstable neurological symptoms within 4 weeks of Cycle 1 Day 1.
6. Major surgery, other than diagnostic surgery, within 2 weeks prior to Cycle 1 Day 1, without complete recovery.
7. Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy.
8. Participant with an established diagnosis of diabetes mellitus Type 1 or not controlled Type 2.
9. Participant has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the trial drugs based on Investigator discretion.
10. Participant has currently documented pneumonitis/interstitial lung disease.
11. Participant has a history of severe cutaneous reaction, such as Stevens-Johnson Syndrome (SJS), Erythema Multiforme (EM), Toxic Epidermal Necrolysis (TEN), or Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS).
12. Other protocol defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | First 28 days (1 cycle) of combination therapy
  Rate of DLTs per dose level
Descriptive statistics of Adverse Events (AEs) | From Cycle 1 Day 1 until 30 days after last trial intervention dose or 30 days after trial completion, whichever comes first, assessed up to 2 years
  Descriptive statistics of Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs; AE severity will be assessed per the NCI CTCAE v 5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From Cycle 1 Day 1 until first documentation of disease progression, the start of new anti-cancer therapy, or death, whichever occurs first, assessed up to 2 years
  Overall confirmed response rate (Complete Response or Partial Response)
Median duration of response | From first documentation of response to first documentation of disease progression, the start of new anti-cancer therapy, or death, whichever occurs first, assessed up to 2 years
  Defined for participants with confirmed objective response as the time from the first documentation of response to the first documentation of disease progression by RECIST v1.1 or to death due to any cause before new anti-cancer treatment, whichever occurs first
Disease control rate (DCR) | From Cycle 1 Day 1 until first documentation of disease progression, the start of new anti-cancer therapy, or death, whichever occurs first, assessed up to 2 years
  Disease control rate (CR + PR + SD)
Median duration of Disease Control | From first documentation of response until first documentation of disease progression, the start of new anti-cancer therapy, or death, whichever occurs first, assessed up to 2 years
  Defined for participants with confirmed objective response as the time in months from the first documentation of response to the first documentation of disease progression by RECIST v1.1 or to death due to any cause before new anti-cancer treatment, whichever occurs first, in patients with confirmed CR/PR
Rate of Stable Disease | From Cycle 1 Day 1 until first documentation of disease progression, the start of new anti-cancer therapy, or death, whichever occurs first, assessed up to 2 years
Median duration of Stable Disease (SD) | From first documentation of response until first documentation of disease progression, the start of new anti-cancer therapy, or death, whichever occurs first, assessed up to 2 years
  Defined as durable SD (>= 12 weeks) by RECIST v1.1
Cmax of tipifarnib and alpelisib when administered in combination | Blood samples will be collected on day 1 and day 2 of Cycle 1 and Cycle 2, and on day 1 of Cycle 3 through Cycle 6. Each cycle is 28 days.
  Peak drug concentration for single dose and multiple dose
Tmax of tipifarnib and alpelisib when administered in combination | Blood samples will be collected on day 1 and day 2 of Cycle 1 and Cycle 2, and on day 1 of Cycle 3 through Cycle 6. Each cycle is 28 days.
  Time to reach peak concentration following drug administration for single dose and multiple dose
AUC(0-last) of tipifarnib and alpelisib when administered in combination | Blood samples will be collected on day 1 and day 2 of Cycle 1 and Cycle 2, and on day 1 of Cycle 3 through Cycle 6. Each cycle is 28 days.
  Area under the concentration-time curve from time zero to time of last measurable concentration for single dose and multiple dose
AUC(tau) of tipifarnib and alpelisib when administered in combination | Blood samples will be collected on day 1 and day 2 of Cycle 1 and Cycle 2, and on day 1 of Cycle 3 through Cycle 6. Each cycle is 28 days.
  Area under the concentration-time curve during a dosage interval for single dose and multiple dose
AUC(0-infinity) of tipifarnib and alpelisib when administered in combination | Blood samples will be collected on day 1 and day 2 of Cycle 1 and Cycle 2, and on day 1 of Cycle 3 through Cycle 6. Each cycle is 28 days.
  Area under the concentration-time curve from time zero to infinity for single dose
CL/F of tipifarnib and alpelisib when administered in combination | Blood samples will be collected on day 1 and day 2 of Cycle 1 and Cycle 2, and on day 1 of Cycle 3 through Cycle 6. Each cycle is 28 days.
  Apparent total clearance of the drug after administration for single dose and multiple dose
Vd/F of tipifarnib and alpelisib when administered in combination | Blood samples will be collected on day 1 and day 2 of Cycle 1 and Cycle 2, and on day 1 of Cycle 3 through Cycle 6. Each cycle is 28 days.
  Apparent volume of distribution after administration for single dose and multiple dose
Half-life of tipifarnib and alpelisib when administered in combination | Blood samples will be collected on day 1 and day 2 of Cycle 1 and Cycle 2, and on day 1 of Cycle 3 through Cycle 6. Each cycle is 28 days.
  Time required for the amount of drug in the body to decrease by half for single dose and multiple dose
Accumulation ratio of tipifarnib and alpelisib when administered in combination | Blood samples will be collected on day 1 and day 2 of Cycle 1 and Cycle 2, and on day 1 of Cycle 3 through Cycle 6. Each cycle is 28 days.
  Ratio of accumulation of a drug after multiple doses compared to a single dose
Progression-free survival (PFS) | From Cycle 1 Day 1 until first documentation of disease progression, the start of new anti-cancer therapy, or death, whichever occurs first, assessed up to 3 years
  Median PFS
Proportion of participants with PFS at 6 months | From Cycle 1 Day 1 until first documentation of disease progression, the start of new anti-cancer therapy, or death, whichever occurs first, assessed up to 6 months
  Proportion of participants alive and without progression at 6 months
Overall Survival (OS) | From Cycle 1 Day 1 until 3 years of treatment or death from any cause, whichever comes first
  Median OS; for patients with no events, OS will be censored at the last known to be alive date
Proportion of patients with OS at 12 months | From Cycle 1 Day 1 until 12 months of treatment or death from any cause, whichever comes first
  For patients with no events, OS will be censored at the last known to be alive date

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Lake Nona DDU (Florida Cancer Specialists), Orlando, Florida
  - University of Maryland School of Medicine (Marlene and Stewart Greenebaum Comprehensive Cancer Center), Baltimore, Maryland
  - Johns Hopkins University School of Medicine (Sidney Kimmel Comprehensive Cancer Center), Baltimore, Maryland
  - Dana-Farber Cancer Institute (Head and Neck Cancer Treatment Center), Boston, Massachusetts
  - Washington University, School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center (Harold C. Simmons Comprehensive Cancer Center), Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin